CLINICAL TRIAL: NCT07335393
Title: Cognition Assessment and REhabilitation in Virtual Reality for Patients With Cancer (CARE-VR4PC)
Brief Title: Cognition Assessment and REhabilitation in Virtual Reality for Patients With Cancer
Acronym: CARE-VR4PC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JING MINGXUE (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor-Investigator, JING MINGXUE, Dr, National University Health System, Singapore
Organization: National University Health System, Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2025-0993; NUSSUG2025 (Other Grant/Funding Number: National University of Singapore Start-up Grant)
Record Dates: First submitted 2025-12-30; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Patients With Cancer
Keywords: Cancer; Virtual Reality; Cognitive Rehabilitation Therapy; Cancer-related cognitive impairment; Quality of Life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: 1. The intervention arm will receive 12 VR-CRT sessions over 4 weeks, with sessions occurring 3 times per week, targeting attention, memory, and executive function.
  2. The control arm will receive standard care only.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-based cognitive rehabilitation therapy (VR-CRT) (Experimental): Intervention Arm
  Interventions: Behavioral: VR-based cognitive rehabilitation therapy (VR-CRT)
- Standard Care only (No Intervention): Control arm

INTERVENTIONS:
Behavioral: VR-based cognitive rehabilitation therapy (VR-CRT) — 12 VR-CRT sessions over 4 weeks, with sessions occurring 3 times per week, targeting attention, memory, and executive function
  Arms: VR-based cognitive rehabilitation therapy (VR-CRT)

SUMMARY:
1. To assess the cognitive function of patients with cancer by leveraging a validated virtual reality (VR)-based cognitive assessment tool.
2. To evaluate the efficacy of VR-based cognitive rehabilitation therapy (VR-CRT) compared to a control group in improving cognitive functions in cancer patients.

Hypothesis

Cancer patients with cancer-related cognitive impairment who receive the VR-CRT program will demonstrate significantly greater improvement in cognitive functions, as measured by the validated VR cognition assessment tool, compared to those who receive standard care, both immediately post-intervention and at 3-month follow-up.

DETAILED DESCRIPTION:
In this prospective, assessor-blinded, randomized controlled study, a total of 64 participants with cancer-related cognitive impairment will be recruited from oncology inpatient wards and outpatient clinics at a tertiary cancer center. 32 participants will be randomized to the intervention arm (VR-based cognitive rehabilitation therapy [VR-CRT]) and 32 participants will be randomized to the control arm (standard care).

The study will consist of a screening period of up to 14 days. Participants who fulfill all inclusion criteria will be consented and recruited during this screening period, constituting Visit 1 (Recruitment). During this visit, the principal investigator (PI) or co-investigator (Co-I) obtaining consent will ensure that the patient meets the following criteria:

For patients where a caregiver may assist with VR setup or monitoring, the study team will ensure that they are the primary caregiver of the patient.

Patient must be comfortable and committed to following directions for VR device usage.

Patient must not have severe cognitive or sensory impairments that preclude safe VR engagement.

After confirmation of the above criteria, the patient will undergo a 1-hour hands-on training session at the cancer center by trained study team members.

A set of training slides titled "VR-CRT User Training Slides" that is adapted from the standard "VR-CRT Instruction Manual" will be utilized for the training session for the patient. After which, a checklist titled "VR Training Checklist" will be completed by both the trainer and patient. This checklist is aimed to ensure that all necessary components of training have been covered by the trainer and also for trainers to indicate confidence of the patient during the training before both trainer and patient sign as a form of training acknowledgement.

Post training, a copy of the standard "VR-CRT Instruction Manual" will be given to the patient. Study team will emphasize to the patient that they can contact the study team at any juncture where they need additional clarifications relating to the device.

Depending on the treatment status at time of screening, the patient will be seen in the inpatient ward or specialist outpatient clinic at day 14 which is considered as Visit 2 (Randomization with allowance + 3 days). Allowance of up to 3 days is given in the event day 14 falls on a weekend/long weekend. Following Visit 2 (Randomization with allowance + 3 days), up to 3 days of habituation for VR device use and tolerability will take place. Participants will be required to engage with the VR device at low levels of immersion to allow conditioning for the habituation period. Because of the nature of the intervention, it may cause some discomfort to the participants, such as mild cybersickness, hence conditioning will increase the tolerability of the treatment for the participants.

Intervention with VR-CRT will take place over 8 weeks either in the inpatient setting of the cancer center or in the home setting, while standard oncology supportive care sessions happening concurrently as per existing clinical treatment protocol. Treatment with VR-CRT will consist of a daily session of 30-45 minutes for 24 sessions over 8 weeks (3 sessions per week). Compliance will be checked by research assistant via telephone or video call interview at regular intervals. One group will be randomized to the standard care (Control) arm and one group will be randomized to the active VR-CRT intervention arm. The standard care (Control) arm will involve routine oncology follow-up and educational resources on cognitive symptom management but no active VR engagement, with assessments conducted in a comparable manner to maintain blinding.

Assessment will be done at the time of recruitment which constitutes as Visit 1 (Recruitment), and again at Visit 3 (Last day of intervention, Week 8 post-intervention with allowance of + 7 days) and Visit 4 (Final follow-up, Week 20 post-intervention with allowance of + 7 days).

Management of adverse events (AEs and SAEs):

At recruitment, patients will be informed to take note and save research coordinator's contact number stated in the informed consent form (ICF). Patients will be reminded to contact research coordinators if patients experience any AE/SAE stated on ICF section 6 from the day of recruitment up to randomization. At randomization it will again be emphasized to patients that they are to continue to monitor for AE/SAE. During the duration of habituation through to the 8-week intervention period, patients are additionally required to report to the study coordinators with regards to any discomfort or issues with the device before proceeding with intervention. During the habituation and the 8-week intervention period, study coordinator will be keeping close contact with the patient by means of messaging apps to ensure compliance to the treatment regime and for AE/SAE reporting.

Patients who are starting the intervention in the inpatient setting will be monitored by the study team for any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* (1) Cancer (both Solid and haematological) patients with documented cognitive impairments. (2) No history of neurological disorders. (3) Ability to use VR technology.

Exclusion Criteria:

* Severe visual or auditory impairments, motion sickness, or conditions interfering with VR use.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
VR Cognition Assessment Tool | From enrollment to Day 90 post-intervention (with allowance of + 7 days).
  Effects of VR-based cognitive rehabilitation therapy (VR-CRT) compared to standard care only (Control) on cognitive function measured objectively using VR Cognition Assessment Tool. Mean change in VR Cognition Assessment Tool from Visit 1 (Recruitment) to Visit 2 (Last day of intervention), and Visit 3 (Final follow-up, Day 90 post-intervention with allowance of + 7 days).
Subjective cognitive function by FACT-Cog | From enrollment to Day 90 post-intervention (with allowance of + 7 days).
  Effects of VR-based cognitive rehabilitation therapy (VR-CRT) compared to standard care only (Control) on subjective cognitive function measured using Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog). Mean change in FACT-Cog from Visit 1 (Recruitment) to Visit 2 (Last day of intervention), and Visit 3 (Final follow-up, Day 90 post-intervention with allowance of + 7 days).

SECONDARY OUTCOMES:
EQ5D-5L | From enrollment to Day 90 post intervention (with allowance of + 7 days).
  Effects of VR-based cognitive rehabilitation therapy (VR-CRT) compared to standard care only (Control) on quality of life (QOL) measured objectively using EQ5D-5L. Mean change in EQ5D-5L from Visit 1 (Recruitment) to Visit 2 (Last day of intervention), and Visit 3 (Final follow-up, Day 90 post intervention with allowance of + 7 days).
Virtual Reality Simulation Sickness Questionnaire (VRSQ) | From enrollment to Day 90 post-intervention (with allowance of + 7 days).
  Effects of VR-based cognitive rehabilitation therapy (VR-CRT) compared to standard care only (Control) on simulation sickness measured objectively using Virtual Reality Simulation Sickness Questionnaire (VRSQ). Mean change in VRSQ from Visit 1 (Recruitment) to Visit 2 (Last day of intervention), and Visit 3 (Final follow-up, Day 90 post-intervention with allowance of + 7 days).
User-friendliness and engagement | From enrollment to Day 90 post-intervention (with allowance of + 7 days).
  Effects of VR-based cognitive rehabilitation therapy (VR-CRT) compared to standard care only (Control) on From enrollment to Day 90 post-intervention (with allowance of + 7 days). assessed using a 9-item scale developed from Makransky and Lilleholt. Mean change in the 9-item scale from Visit 1 (Recruitment) to Visit 2 (Last day of intervention), and Visit 3 (Final follow-up, Day 90 post-intervention with allowance of + 7 days).
Treatment satisfaction by VAS | From enrollment to Day 90 post-intervention (with allowance of + 7 days)
  Effects of VR-based cognitive rehabilitation therapy (VR-CRT) compared to standard care only (Control) on treatment satisfaction measured using Visual Analog Scale (VAS). Mean change in VAS from Visit 1 (Recruitment) to Visit 2 (Last day of intervention), and Visit 3 (Final follow-up, Day 90 post-intervention with allowance of + 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Yingchun Zeng, Principal Investigator — National University of Singapore

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Analytic Code
Time Frame: Beginning 6 months and ending 1 years after the publication of results
Access Criteria: Analyses that qualify for data sharing: meta-analysis Data sharing agreement needs to be signed. Applicant can email the study's Principal Investigator to submit request.

REFERENCES:
- [Result] Zeng Y, Guan Q, Su Y, Huang Q, Zhao J, Wu M, Guo Q, Lyu Q, Zhuang Y, Cheng AS. A self-administered immersive virtual reality tool for assessing cognitive impairment in patients with cancer. Asia Pac J Oncol Nurs. 2023 Feb 28;10(3):100205. doi: 10.1016/j.apjon.2023.100205. eCollection 2023 Mar. PMID 37012969
- [Result] Zeng Y, Zeng L, Cheng ASK, Wei X, Wang B, Jiang J, Zhou J. The use of immersive virtual reality for cancer-related cognitive impairment assessment and rehabilitation: A clinical feasibility study. Asia Pac J Oncol Nurs. 2022 May 17;9(12):100079. doi: 10.1016/j.apjon.2022.100079. eCollection 2022 Dec. PMID 36276883